CLINICAL TRIAL: NCT02375503
Title: Efficacy of a Once Daily Calcium and Vitamin D Fortified Food Product to Improve Bone Microarchitecture in Response to Army Basic Combat Training
Brief Title: Efficacy of a Once Daily Calcium and Vitamin D Fortified Food Product to Improve Bone Microarchitecture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-07-HC
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Bone Alteration; Dietary Modification
Keywords: Calcium; Vitamin D; Parathyroid Hormone; Bone; Microarchitecture
MeSH Terms: interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium/Vitamin D (Experimental): Dietary supplement distributed and consumed as one calcium and vitamin D fortified snack bar per day
  Interventions: Dietary Supplement: Calcium/Vitamin D
- Placebo (Placebo Comparator): Placebo distributed and consumed as one isocaloric, unfortified snack bar per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Calcium/Vitamin D — Daily, calcium and vitamin D fortified snack bar
  Arms: Calcium/Vitamin D
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this randomized, double-blind, placebo controlled trial is to determine the efficacy of a once per day calcium (1000mg) and vitamin D (1000IU) fortified food product on bone turnover markers, including parathyroid hormone (PTH) and microarchitecture during Army basic military training (BCT). The investigators hypothesize that consumption of a once daily calcium and vitamin D fortified food product will stabilize PTH and contribute to improved bone microarchitecture compared to placebo. The results will determine the efficacy of daily supplementation with calcium and vitamin D on bone turnover markers as well as provide novel data regarding microarchitectural changes during BCT as assessed by high resolution peripheral computed tomography (HRpQCT) scanning.

DETAILED DESCRIPTION:
Stress fractures may affect up to 2-5% of male and 8-21% of female Soldiers during training, resulting in attrition in up to 60% of affected personnel. A recent report indicates that supplemental calcium (2000mg) and vitamin D (800-1000IU) stabilizes PTH, increases tibia volumetric bone mineral density in male and female recruits undergoing Army BCT, and reduces stress fracture incidence by up to 20% in female Nacy recruits. Bone macroarchitecture has been measured in response to basic training however, the resolution of standard peripheral quantitative computed tomography (pQCT) is insufficient for assessment of microarchitectural changes, which may underlie the pathophysiology of stress fracture. With the use of HRpQCT this study will allow the investigators to evaluate microarchitectural changes within the bone tissue and assess the efficacy of a moderate daily dose of calcium and vitamin D to support bone health during BCT.

ELIGIBILITY:
Inclusion Criteria:

* Female or male US Army recruits beginning Army basic combat training at Fort Jackson, South Carolina

Exclusion Criteria:

* Pregnant or breastfeeding
* History of kidney stones or kidney disease
* History of amenorrhea
* History or endocrine disorders
* History of bone modifying disorders
* Currently taking, or have taken glucocorticoid drugs in the 2 years prior to study participation
* Currently diagnosed as anemic by healthcare professional
* Those allergic to any component of the snack bar

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Bone Turnover Markers | 8-10 weeks
  Participants will have a pre- and post- BCT blood draw

SECONDARY OUTCOMES:
Bone Microarchitecture | 8-10 weeks
  Participants will receive a bone scan pre- and post- BCT in order to determine changes in bone microarchitecture

CONTACTS AND LOCATIONS:
Overall Officials: Erin Gaffney-Stomberg, Ph.D., R.D., Principal Investigator — U.S. Army Research Institute of Environmental Medicine
Locations (1):
- Fort Jackson, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lutz LJ, Gaffney-Stomberg E, Karl JP, Hughes JM, Guerriere KI, McClung JP. Dietary Intake in Relation to Military Dietary Reference Values During Army Basic Combat Training; a Multi-center, Cross-sectional Study. Mil Med. 2019 Mar 1;184(3-4):e223-e230. doi: 10.1093/milmed/usy153. PMID 29982620